CLINICAL TRIAL: NCT03790670
Title: Safety, Tolerability and Biomarker Assessments of Leukine (Sargramostim) During Extended Timed Treatment for Parkinson's Disease: A Phase I Pilot Study
Brief Title: Biomarker Assessments of Leukine During Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0839-18-FB
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leukine Treatment (Experimental): 36 month regimen of Leukine administered as a weight-based dose at 3 µg/kg/day for 5 days (week), followed by a 2-day holiday (weekend)
  Interventions: Drug: sargramostim

INTERVENTIONS:
Drug: sargramostim — Recombinant human GM-CSF produced by recombinant DNA technology using a yeast (S. cerevisiae) expression system
  Other Names: Leukine

SUMMARY:
First, the investigators will determine the safety of a 36 month regimen of Leukine administered as a weight-based dose at 3 µg/kg/day for 5 days (week), followed by a 2-day holiday (weekend). This 36 month (n=10) pilot study will extend the prior 2 month observation tests towards the goal of assessing the safety of Leukine for treatment of Parkinson's disease (PD). Clinical signs and symptoms will be measured by personal well-being, physical, and neurological examinations (UPDRS Parts I, II, III, and IV assessments) and blood tests (CBC with differential, total T cell count, and a comprehensive metabolic sera panel). Second, we will assess regimen tolerability administered in a dose reduction, from 6 µg/kg/day without interruption, to 3 µg/kg/day with 2 day drug holidays. The investigators will examine over a time of 36 months, effects of treatment on defined adaptive immune deficits in PD as measured by analysis of peripheral blood mononuclear cells collected before, during, and after cessation of Leukine administration. Individual T cell parameters will be assessed and will include links between T cell function and subset analyses and clinical neurological signs and symptoms. In addition, the functional stability of the immune deficits will be assess in PD by examining T cell subsets in PD patients in this study against prior results. The investigators will also determine whether the immune deficits of PD are consistent during baseline data collection, and the potential Leukine-induced motor control and mobility improvements will be determined by UPDRS part I, II, III, and IV scores off treatment and on treatment.

DETAILED DESCRIPTION:
Primary Objectives: There are three study goals. First, the investigators will determine the safety of a 36 month regimen of Leukine administered as a weight-based dose at 3 µg/kg/day for 5 days (week), followed by a 2-day holiday (weekend). This 36 month (n=10) pilot study will extend the prior 2 month observation tests towards the goal of assessing the safety of Leukine for treatment of Parkinson's disease (PD). Clinical signs and symptoms will be measured by personal well-being, physical, and neurological examinations (UPDRS Parts I, II, III, and IV assessments) and blood tests (CBC with differential, total T cell count, and a comprehensive metabolic sera panel). Second, the investigators will assess regimen tolerability administered in a dose reduction, from 6 µg/kg/day without interruption, to 3 µg/kg/day with 2 day drug holidays. The lowered dose was chosen based on known tolerability and parallel-linked immune reconstitution seen in cancer-associated disease treatments. Due to fragility of the patient population and prior recorded adverse events the proposed dose reductions are justified.

Secondary Objectives:

Over a course of 36 months, the effects of treatment on defined adaptive immune deficits in PD as measured by analysis of peripheral blood mononuclear cells collected before, during, and after cessation of Leukine administration will be examined. Individual T cell parameters that include links between T cell function and subset analyses and clinical neurological signs and symptoms will be examined. These immune parameters will be serially examined as they may contribute to the immune deficits in PD. Thus, timed analyses of changes in T cell phenotypes and/or function will be completed. In addition, the investigators will assess the functional stability of the immune deficits in PD and will determine whether the immune deficits of PD are consistent during baseline data collection. The potential Leukine-induced motor control and mobility improvements will be determined by assessing UPDRS part I, II, III, and IV scores off treatment and on treatment. Specifically, over the course of this six-month treatment study, various biomarkers will be assessed including: T cell markers of immune activation, DNA methylation status, and B cell and bone marrow progenitor cell markers. We hope to uncover the time course of Treg induction, as well as link the pharmacokinetics of Leukine treatment (not previously recorded) to changes in specific biomarkers. Additionally, changes in the humoral response following extended Leukine treatment will be assessed by measuring the presence of antibodies against Leukine and alterations in B cell frequencies.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of bradykinesia and 1 or both of the following: rest tremor and/or rigidity
2. Asymmetric onset of clinical signs
3. Progressive motor symptoms
4. Age at onset 35-85 years
5. Duration of PD symptoms of at least 3 years
6. Female subjects must be either:

   1. Not pregnant, not breastfeeding, and not planning on becoming pregnant during the study;
   2. Not of childbearing potential, defined as one who has been postmenopausal for at least 1 year and with follicle stimulating hormone (FSH) levels in the laboratory defined postmenopausal range, or has been surgically sterilized, or has had a hysterectomy at least 3 months prior to the start of this trial; or
   3. If of childbearing potential, must agree to use an effective method of avoiding pregnancy to the end of the trial and must have a negative serum beta-human chorionic gonadotropin (β-HCG) test. Effective methods of avoiding pregnancy are contraceptive methods used consistently and correctly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide, or cervical cap), abstinence, or a sterile sexual partner.
7. Must be stage 4 or less according to the Hoehn and Yahr scale

Exclusion Criteria:

1. Atypical features indicative of a Parkinson-Plus disorder (Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD)) including cerebellar signs, supranuclear gaze palsy, apraxia and other cortical signs, or prominent autonomic failure
2. Neuroleptic treatment at time of onset of parkinsonism
3. Active treatment with a neuroleptic at time of study entry
4. History of repeated strokes with stepwise progression of parkinsonism
5. History of repeated head injury
6. History of definite encephalitis
7. More than one blood relative diagnosed with PD
8. Prominent gait imbalance early in the course (< 5 years)
9. Mini-mental state examination score <26
10. Hematological malignancy or coagulopathy
11. Abnormal blood analyses: hematocrit <30; WBC>11.5; clinically significant laboratory data (e.g. alanine aminotransferase [ALT] or aspartate aminotransferase [AST] 3x the upper limit of normal [ULN]), or any abnormal laboratory value that could interfere with the assessment of safety in the judgment of the investigator; significant abnormalities on the clinical examination, vital signs, and clinical chemistry or hematology results (excluding findings of Parkinson's disease), that may interfere with the study or present a safety risk for the subject as judged by the clinical investigator charged in the care of study participants
12. Serious medical illness or co-morbidity that may interfere with participation in the study
13. Brain surgery for parkinsonism (DBS, cell implantation, gene therapy)
14. History of an autoimmune disorder or systemic inflammatory disorder deemed significant by physician
15. Immunostimulatory or immunosuppressive treatment (including amphet-amines or systemic corticosteroids) within 90 days
16. Exclusively unilateral parkinsonism for longer than 3 years
17. Known hypersensitivity to GM-CSF, yeast-derived products
18. Current lithium treatment
19. Individuals with current diagnoses of alcohol or substance abuse/dependence
20. Anyone who is not appropriate for participation in this research protocol as deemed by the principal or co-investigator
21. Anyone who has previously been treated with GM-CSF as an immunomodulatory therapy
22. Anyone with poor venous access

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Associated Adverse Events | monthly during the course of treatment, up to 36 months, followed by 1 month drug cessation
  The safety of Leukine administration in PD will be examined by documenting abnormal results from CBC with differential, total T cell count, or comprehensive metabolic panel analyses; abnormal physical and or neurological exam findings; abnormal levels of antibodies to GM-CSF; clinically increasing Unified Parkinson's disease Rating Scale (UPDRS) part I, II, III, and IV scores as determined by the examining physician; and other adverse events. These safety assessments will be made every four weeks.

SECONDARY OUTCOMES:
Determination of Immune Cell Phenotype | 36 months of treatment, followed by 1 month drug cessation
  Measurements will include change in CD45RO+ or FAS+ frequencies in CD4+ T cells; change in CD31+ frequencies in CD4+ T cells, Teff or Treg subsets; change in ItgB7+ frequencies in CD4+ T cells or the Teff subset; change in ItgB4B7+ frequencies in CD4+ T cells or the Treg subset; change in CD27+ frequencies in CD4+ T cells, Teff or Treg subsets, change in CCR7+ frequencies in CD4+ T cells, Teff or Treg subsets; change in FoxP3+ frequencies in CD4+ T cells, Teff or Treg subsets; change in CD34, CD117, or CD135 levels; change in DNA methylation status. The measurements will be combined to determine overall changes in immune cell frequency and T cell subset phenotype both on and off treatment.
Determination of Immune Cell Number | 36 months of treatment, followed by 1 month drug cessation
  Measurements will include changes in levels of lymphocytes or CD4+ T cells, as well as T cell, B cell, and bone marrow progenitor subsets.
Determination of Immune Cell Function | 36 months of treatment, followed by 1 month drug cessation
  Measurements will include changes in T cell function via proliferation and suppression assays and/or changes in B cell function via antibody production assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gendelman, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gendelman HE, Zhang Y, Santamaria P, Olson KE, Schutt CR, Bhatti D, Shetty BLD, Lu Y, Estes KA, Standaert DG, Heinrichs-Graham E, Larson L, Meza JL, Follett M, Forsberg E, Siuzdak G, Wilson TW, Peterson C, Mosley RL. Evaluation of the safety and immunomodulatory effects of sargramostim in a randomized, double-blind phase 1 clinical Parkinson's disease trial. NPJ Parkinsons Dis. 2017 Mar 23;3:10. doi: 10.1038/s41531-017-0013-5. eCollection 2017. PMID 28649610
- [Background] Saunders JA, Estes KA, Kosloski LM, Allen HE, Dempsey KM, Torres-Russotto DR, Meza JL, Santamaria PM, Bertoni JM, Murman DL, Ali HH, Standaert DG, Mosley RL, Gendelman HE. CD4+ regulatory and effector/memory T cell subsets profile motor dysfunction in Parkinson's disease. J Neuroimmune Pharmacol. 2012 Dec;7(4):927-38. doi: 10.1007/s11481-012-9402-z. Epub 2012 Oct 11. PMID 23054369
- [Background] Kosloski LM, Kosmacek EA, Olson KE, Mosley RL, Gendelman HE. GM-CSF induces neuroprotective and anti-inflammatory responses in 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine intoxicated mice. J Neuroimmunol. 2013 Dec 15;265(1-2):1-10. doi: 10.1016/j.jneuroim.2013.10.009. Epub 2013 Oct 29. PMID 24210793
- [Derived] Olson KE, Abdelmoaty MM, Namminga KL, Lu Y, Obaro H, Santamaria P, Mosley RL, Gendelman HE. An open-label multiyear study of sargramostim-treated Parkinson's disease patients examining drug safety, tolerability, and immune biomarkers from limited case numbers. Transl Neurodegener. 2023 May 22;12(1):26. doi: 10.1186/s40035-023-00361-1. PMID 37217980
- [Derived] Olson KE, Namminga KL, Lu Y, Schwab AD, Thurston MJ, Abdelmoaty MM, Kumar V, Wojtkiewicz M, Obaro H, Santamaria P, Mosley RL, Gendelman HE. Safety, tolerability, and immune-biomarker profiling for year-long sargramostim treatment of Parkinson's disease. EBioMedicine. 2021 May;67:103380. doi: 10.1016/j.ebiom.2021.103380. Epub 2021 May 14. PMID 34000620

DOCUMENTS (1):
  • Informed Consent Form: Informed Consent Form rev1 (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03790670/ICF_000.pdf